CLINICAL TRIAL: NCT01197508
Title: A Multicenter, Randomized, Double-Blind Parallel Group Placebo-Controlled Phase III, Efficacy and Safety Study of 3 Fixed Dose Groups of TC-5214 (S-mecamylamine) as an Adjunct to an Antidepressants in Patients With Major Depressive Disorder Who Exhibit an Inadequate Response to Antidepressant Therapy
Brief Title: A Study to Assess the Efficacy and Safety of TC-5214 as an Adjunct Therapy in Patients With Major Depressive Disorder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4130C00005
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2012-10-29 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-03

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder, MDD, Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 0.1 mg BID TC-5214 (Experimental): Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + TC-5214, 0.1 mg BID
  Interventions: Drug: TC-5214
- 1 mg BID TC-5214 (Experimental): Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + TC-5214, 1 mg BID
  Interventions: Drug: TC-5214
- 4 mg BID TC-5214 (Experimental): Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + TC-5214, 4 mg BID
  Interventions: Drug: TC-5214
- Placebo (Placebo Comparator): Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + Placebo BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TC-5214 — Twice daily for 8 weeks.
  Arms: 0.1 mg BID TC-5214; 1 mg BID TC-5214; 4 mg BID TC-5214
Drug: Placebo — Twice daily for 8 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if TC-5214 or placebo (a tablet that looks like a medicine tablet or capsule, but contains no active medicine) is safe and effective when taken together with another antidepressant.

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-Blind Parallel Group Placebo-Controlled Phase III, Efficacy and Safety Study of 3 Fixed Dose Groups of TC-5214 (S-mecamylamine) as an Adjunct to an Antidepressants in Patients with Major Depressive Disorder Who Exhibit an Inadequate Response to Antidepressant Therapy

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent before initiation of any study-related procedures.
* The patient must have a clinical diagnosis of major depressive disorder (MDD) with inadequate response to no more than one antidepressant.
* Outpatient status at enrollment and randomization.

Exclusion Criteria:

* Patients with a lifetime history of bipolar disorder, psychotic disorder or post-traumatic stress disorder.
* Patients with a history of suicide attempts in the past year and/or seen by the investigator as having a significant history of risk of suicide or homicide.
* History of renal insufficiency or impairment or conditions that could affect absorption or metabolism of investigational product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Actual)
Dates: Start 2010-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans A Eriksson, MD,PhD, MBA, Study Director — AstraZeneca R&D; Hans-Jürgen Möller, Prof. Dr., Principal Investigator — University Hospital München
Locations (87):
- Argentina (4):
  - Research Site, Buenos Aires, Buenos Aires F.D.
  - Research Site, Mendoza, Mendoza Province
  - Research Site, Ciudad Autonoma Bs As, Cba
  - Research Site, Dublin
- Research Site, Rio de Janeiro, Rio de Janeiro, Brazil
- Bulgaria (2):
  - Research Site, Novi Iskar
  - Research Site, Rousse
- Chile (3):
  - Research Site, Santiago, Chile
  - Research Site, Antofagasta
  - Research Site, Providencia Santiago
- Colombia (4):
  - Research Site, Bello, Antioquia
  - Research Site, Bogota, Cundinamarca
  - Research Site, Pereira, Risaralda Department
  - Research Site, Cali, Valle del Cauca Department
- Research Site, Rijeka, Croatia
- France (13):
  - Research Site, Bully-les-Mines
  - Research Site, Caen
  - Research Site, Cherbourg
  - Research Site, Colmar
  - Research Site, Dole
  - Research Site, Douai
  - Research Site, Élancourt
  - Research Site, Montpellier
  - Research Site, Sartrouville
  - Research Site, Strasbourg
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tours
- Germany (6):
  - Research Site, Hüttenberg, Hesse
  - Research Site, Bad Homburg
  - Research Site, Bielefeld
  - Research Site, Gelsenkirchen
  - Research Site, Schwerin
  - Research Site, Siegen
- Hungary (3):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Győr
- Poland (5):
  - Research Site, Bydgoszcz, Poland
  - Research Site, Bialystok
  - Research Site, Leszno
  - Research Site, Lublin
  - Research Site, Torun
- Romania (7):
  - Research Site, Arad
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Focşani
  - Research Site, Oradea
  - Research Site, Timișoara
- Russia (8):
  - Research Site, Arkhangelsk
  - Research Site, Chita
  - Research Site, Novosibirsk
  - Research Site, Petrozavodsk
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
  - Research Site, Voronezh
  - Research Site, Yekaterinburg
- Serbia (2):
  - Research Site, Kragujevac, Serbia and Montenegro
  - Research Site, Niš
- Slovakia (7):
  - Research Site, Banská Štiavnica
  - Research Site, Bratislava
  - Research Site, Levice
  - Research Site, Prešov
  - Research Site, Rimavská Sobota
  - Research Site, Svidník
  - Research Site, Trenčín
- South Africa (8):
  - Research Site, Bloemfontein, Free State
  - Research Site, Vereeniging, Free State
  - Research Site, Cape Town, Western Cape
  - Research Site, Centurion
  - Research Site, Durban
  - Research Site, George
  - Research Site, Paarl
  - Research Site, Port Elizabeth
- Spain (3):
  - Research Site, Alcalá de Henares, Madrid
  - Research Site, Coslada, Madrid
  - Research Site, Langreo, Principality of Asturias
- Ukraine (10):
  - Research Site, Kharkiv, Ukraine
  - Research Site, Simferpool, Ukraine
  - Research Site, Vinnytsia, Ukraine
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kherson
  - Research Site, Kiev
  - Research Site, Lviv
  - Research Site, Poltava
  - Research Site, Ternopil

REFERENCES:
- [Derived] Moller HJ, Demyttenaere K, Olausson B, Szamosi J, Wilson E, Hosford D, Dunbar G, Tummala R, Eriksson H. Two Phase III randomised double-blind studies of fixed-dose TC-5214 (dexmecamylamine) adjunct to ongoing antidepressant therapy in patients with major depressive disorder and an inadequate response to prior antidepressant therapy. World J Biol Psychiatry. 2015 Oct;16(7):483-501. doi: 10.3109/15622975.2014.989261. Epub 2015 Jan 20. PMID 25602163
- See also: CSR-D4130C00005.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=336&filename=CSR-D4130C00005.pdf
- See also: D4130C00005/Clinical Study Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=336&filename=D4130C00005_Revised_CSP_1_redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in Europe, South Africa, and Latin America between 1 September 2010 and 30 January 2012.
Pre-assignment Details: The study had an up to 21-day screening/washout period, and an 8-week prospective open-label antidepressant treatment (ADT) period to identify the target patient population of inadequate responders to ADT (<50% reduction in HAMD-17 total score during the prospective open-label ADT period, a HAMD-17 total score of ≥16 and a CGI-S score ≥4).
Period: Overall Study
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Started | 174 | 174 | 174 | 174
Received Treatment | 174 | 174 | 171 | 174
Completed | 151 | 144 | 125 | 158
Not Completed | 23 | 30 | 49 | 16
Not completed — Withdrawal by Subject | 8 | 7 | 15 | 4
Not completed — Eligiblity criteria not fulfilled | 0 | 0 | 2 | 0
Not completed — Adverse Event | 10 | 13 | 23 | 3
Not completed — Severe non-compliance to protocol | 0 | 3 | 1 | 3
Not completed — Condition under investigation worsened | 1 | 1 | 1 | 1
Not completed — Lack of Efficacy | 1 | 2 | 2 | 1
Not completed — Study-specific withdrawal criteria | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 1 | 1 | 2 | 0
Not completed — Other | 2 | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo | Total
Number analyzed (Participants) | 174 | 174 | 174 | 174 | 696
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (10.66) | 45.0 (11.72) | 45.6 (10.72) | 45.8 (11.75) | 45.6 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 125 | 117 | 129 | 498
  Male | 47 | 49 | 57 | 45 | 198
Race/Ethnicity, Customized [Number; unit: participants]
  White | 161 | 156 | 157 | 158 | 632
  Black or African American | 2 | 3 | 1 | 2 | 8
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Other | 11 | 13 | 16 | 13 | 53
Hamilton Rating Scale for Depression-17 items (HAMD-17) total score at randomization [Mean (Standard Deviation); unit: Scores on a scale] — A 17-item, clinician-rated scale that assesses depressive symptoms. The HAMD-17 consists of 17 symptoms, each of which is rated from 0 to 2 or 0 to 4, where 0 is none/absent. The HAMD-17 total score is calculated as the sum of the 17 individual symptom scores; the total score can range from 0 to 52. Higher HAMD-17 scores indicate more severe depression.
  Scores on a scale | 21.49 (3.587) | 20.98 (3.182) | 21.50 (3.674) | 21.26 (3.614) | 21.30 (3.517)
Montgomery-Asberg Depression Rating Scale (MADRS) total score at randomization [Mean (Standard Deviation); unit: Scores on a scale] — A 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
  Scores on a scale | 24.69 (5.086) | 24.67 (5.389) | 25.03 (5.137) | 24.11 (4.992) | 24.62 (5.152)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score From Randomization to End of Treatment.
Description: A 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: Modified intent-to-treat analysis set including all randomized patients who received at least 1 dose of investigational product (TC-5214 or placebo) and who had a randomization and at least 1 post-randomization MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 173 | 174 | 170 | 174
units on a scale | -11.6 (0.65) | -12.2 (0.66) | -12.2 (0.69) | -12.7 (0.65)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; Mixed model repeated measures (MMRM) includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization MADRS total score as a covariate. Treatment, visit and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 1.000, MMRM — The adjusted p-value protects the overall family-wise error rate by taking into account the multiple comparisons between the TC-5214 doses for both the primary efficacy variable (MADRS) and the key secondary efficacy variable (SDS); LS mean = 1.1, 95% CI 2-sided [-0.53 to 2.79], Standard Error of Mean 0.84
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.000, MMRM; LS mean = 0.5, 95% CI 2-sided [-1.22 to 2.13], Standard Error of Mean 0.85
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.000, MMRM; LS mean = 0.5, 95% CI 2-sided [-1.21 to 2.22], Standard Error of Mean 0.88

2. Secondary Outcome: Response in Depressive Symptoms of Major Depressive Disorder (MDD), Defined as a ≥50% Reduction From Randomization (Week 8) in MADRS Total Score at End of Treatment (Week 16)
Description: The percentage of patients with a ≥50% reduction from randomization (Week 8) in MADRS total score at end of treatment (Week 16) was calculated.
  MADRS is 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Number; unit: percentage of participants analyzed
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 173 | 174 | 170 | 174
percentage of participants analyzed | 48.6 | 51.1 | 41.2 | 54.0
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; Logistic regression model including treatment and pooled center as fixed effects and the randomization MADRS total score as a covariate; Test type: Superiority or Other; p = 0.144, Regression, Logistic; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.45 to 1.12], Standard Error of Mean 0.17 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.203, Regression, Logistic; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.47 to 1.17], Standard Error of Mean 0.17 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.32 to 0.82], Standard Error of Mean 0.12 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214

3. Secondary Outcome: Remission in Depressive Symptoms of MDD, Defined as MADRS Total Score of ≤8 at End of Treatment (Week 16)
Description: The percentage of patients with a MADRS total score of ≤8 at end of treatment (Week 16) was calculated.
  MADRS is 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants analyzed
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 173 | 174 | 170 | 174
percentage of participants analyzed | 37.0 | 35.1 | 30.0 | 39.1
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.636, Regression, Logistic; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.54 to 1.45], Standard Error of Mean 0.22 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.215, Regression, Logistic; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.44 to 1.20], Standard Error of Mean 0.19 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.034, Regression, Logistic; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.35 to 0.96], Standard Error of Mean 0.15 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214

4. Secondary Outcome: Early and Sustained Response, Defined as a ≥50% Reduction From Randomization (Week 8) in MADRS Total Score and a MADRS Total Score of ≤12 at Week 10, Week 12, Week 14, and End of Treatment (Week 16)
Description: The percentage of patients with a ≥50% reduction from randomization (Week 8) in MADRS total score and a MADRS total score of ≤12 at Week 10, Week 12, Week 14, and end of treatment (Week 16) was calculated.
  MADRS is 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Randomization (Week 8) to end of treatment (Week 16); Week 10, Week 12, Week 14, and Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants analyzed
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 173 | 173 | 166 | 173
percentage of participants analyzed | 7.5 | 8.1 | 9.6 | 9.2
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.711, Regression, Logistic; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.36 to 1.99], Standard Error of Mean 0.37 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.594, Regression, Logistic; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.34 to 1.85], Standard Error of Mean 0.34 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.749, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.50 to 2.65], Standard Error of Mean 0.49 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214

5. Secondary Outcome: Sustained Response, Defined as a ≥50% Reduction From Randomization (Week 8) in MADRS Total Score and a MADRS Total Score of ≤12 at Week 12, Week 14, and End of Treatment (Week 16)
Description: The percentage of patients with a ≥50% reduction from randomization (Week 8) in MADRS total score and a MADRS total score of ≤12 at Week 12, Week 14, and end of treatment (Week 16) was calculated.
  MADRS is 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Randomization (Week 8) to end of treatment (Week 16); Week 12, Week 14, and Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of patients analyzed
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 170 | 171 | 163 | 173
percentage of patients analyzed | 14.7 | 19.3 | 15.3 | 23.7
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.037, Regression, Logistic; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.28 to 0.96], Standard Error of Mean 0.16 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.222, Regression, Logistic; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.38 to 1.25], Standard Error of Mean 0.21 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.042, Regression, Logistic; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.28 to 0.98], Standard Error of Mean 0.17 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214

6. Secondary Outcome: Sustained Remission, Defined as a MADRS Total Score of ≤8 at Week 12, Week 14, and End of Treatment (Week 16)
Description: The percentage of patients with a MADRS total score of ≤8 at Week 12, Week 14, and end of treatment (Week 16)was calculated.
  MADRS is 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Week 12, Week 14, Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants analyzed
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 170 | 172 | 163 | 173
percentage of participants analyzed | 10.6 | 10.5 | 8.0 | 12.1
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.913, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.48 to 2.27], Standard Error of Mean 0.41 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.841, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.42 to 2.01], Standard Error of Mean 0.37 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.239, Regression, Logistic; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.26 to 1.39], Standard Error of Mean 0.26 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214

7. Secondary Outcome: Change in Depressive Symptoms From Randomization (Week 8) to End of Treatment (Week 16) as Measured by Hamilton Rating Scale for Depression-17 Items (HAMD-17) Total Score
Description: A 17-item, clinician-rated scale that assesses depressive symptoms. The HAMD-17 consists of 17 symptoms, each of which is rated from 0 to 2 or 0 to 4, where 0 is none/absent. The HAMD-17 total score is calculated as the sum of the 17 individual symptom scores; the total score can range from 0 to 52. Higher HAMD-17 scores indicate more severe depression.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 165 | 161 | 162 | 170
units on a scale | -10.07 (0.597) | -10.21 (0.603) | -9.07 (0.597) | -11.16 (0.592)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; Analysis of covariance (ANCOVA) with randomization HAMD-17 total score as covariate, treatment as a fixed effect and pooled center as a random effect; Test type: Superiority or Other; p = 0.120, ANCOVA; LS mean = 1.10, 95% CI 2-sided [-0.288 to 2.481], Standard Error of Mean 0.705
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.184, ANCOVA; LS mean = 0.95, 95% CI 2-sided [-0.452 to 2.354], Standard Error of Mean 0.715
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.003, ANCOVA; LS mean = 2.09, 95% CI 2-sided [0.692 to 3.484], Standard Error of Mean 0.711

8. Secondary Outcome: Change in the Clinician-rated Global Outcome of Severity as Measured by the Clinical Global Impression-Severity (CGI-S) Score From Randomization (Week 8) to End of Treatment (Week 16)
Description: A 3-part, clinician-administered scale that rates the improvement or worsening of the patient's illness from randomization (baseline). Each item is scored on a 1 to 7 scale. Higher CGI-S scores indicate greater illness severity.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 173 | 174 | 170 | 174
units on a scale | -1.5 (0.09) | -1.6 (0.09) | -1.7 (0.10) | -1.7 (0.09)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit, and treatment by visit interaction as explanatory variables and the randomization CGI-S total score as a covariate. Treatment, visit, and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.131, MMRM; LS mean = 0.2, 95% CI [-0.05 to 0.42], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.551, MMRM; LS mean = 0.1, 95% CI 2-sided [-0.17 to 0.31], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.645, MMRM; LS mean = 0.1, 95% CI 2-sided [-0.19 to 0.30], Standard Error of Mean 0.12

9. Secondary Outcome: Response in the Clinical Global Impression-Improvement (CGI-I) Defined as CGI-I Rating of "Very Much Improved" or "Much Improved" From Randomization (Week 8) to End of Treatment (Week 16)
Description: A 3-part, clinician-administered scale that rates the improvement or worsening of the patient's illness from randomization (baseline). Each item is scored on a 1 to 7 scale. CGI-I scores >4 indicate worsening, while scores <4 indicate improvement.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Number; unit: percentage of participants analyzed
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 173 | 174 | 170 | 174
percentage of participants analyzed | 59.5 | 62.1 | 58.8 | 67.8
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; Logistic regression model including treatment and pooled center as fixed effects and the randomization Clinical Global Impression Severity (CGI-S) as a covariate; Test type: Superiority or Other; p = 0.046, Regression, Logistic; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.38 to 0.99], Standard Error of Mean 0.15 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.051, Regression, Logistic; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.38 to 1.00], Standard Error of Mean 0.15 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.040, Regression, Logistic; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.37 to 0.98], Standard Error of Mean 0.15 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214

10. Secondary Outcome: Change in Hamilton Anxiety Scale (HAM-A) Total Score From Randomization (Week 8) to End of Treatment (Week 16)
Description: A 14-item clinician-administered scale for the evaluation of anxiety symptoms. Each HAM-A item is rated on a 0 to 4 scale. Higher HAM-A scores indicate higher levels of anxiety.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 166 | 161 | 161 | 170
units on a scale | -8.5 (0.58) | -8.6 (0.59) | -8.1 (0.58) | -9.3 (0.58)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; An analysis of covariance (ANCOVA) with randomization HAM-A total score as covariate, treatment as a fixed effect and pooled center as a random effect; Test type: Superiority or Other; p = 0.273, ANCOVA; LS mean = 0.7, 95% CI 2-sided [-0.58 to 2.03], Standard Error of Mean 0.66
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.315, ANCOVA; LS mean = 0.7, 95% CI 2-sided [-0.65 to 2.00], Standard Error of Mean 0.67
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.078, ANCOVA; LS mean = 1.2, 95% CI 2-sided [-0.13 to 2.51], Standard Error of Mean 0.67

11. Secondary Outcome: Change in MADRS Total Score From Randomization (Week 8) to Week 9
Description: as for outcome 1
Time Frame: Randomization (Week 8) to Week 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 167 | 162 | 164 | 168
units on a scale | -3.0 (0.42) | -3.0 (0.43) | -2.6 (0.42) | -3.2 (0.42)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization MADRS total score as a covariate. Treatment, visit and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.590, MMRM; LS mean = 0.3, 95% CI 2-sided [-0.68 to 1.19], Standard Error of Mean 0.47
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.679, MMRM; LS mean = 0.2, 95% CI 2-sided [-0.74 to 1.14], Standard Error of Mean 0.48
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.215, MMRM; LS mean = 0.6, 95% CI 2-sided [-0.35 to 1.53], Standard Error of Mean 0.48

12. Secondary Outcome: Change in MADRS Total Score From Randomization (Week 8) to Week 10
Description: as for outcome 1
Time Frame: Randomization (Week 8) to Week 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 170 | 166 | 157 | 171
units on a scale | -4.8 (0.50) | -5.9 (0.50) | -5.0 (0.51) | -6.0 (0.50)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.052, MMRM; LS mean = 1.2, 95% CI 2-sided [-0.01 to 2.38], Standard Error of Mean 0.61
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.874, MMRM; LS mean = 0.1, 95% CI 2-sided [-1.11 to 1.30], Standard Error of Mean 0.61
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.099, MMRM; LS mean = 1.0, 95% CI 2-sided [-0.19 to 2.24], Standard Error of Mean 0.62

13. Secondary Outcome: Change in MADRS Total Score From Randomization (Week 8) to Week 12
Description: as for outcome 1
Time Frame: Randomization (Week 8) to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 163 | 157 | 144 | 166
units on a scale | -8.1 (0.55) | -8.5 (0.56) | -7.8 (0.57) | -8.7 (0.55)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.394, MMRM; LS mean = 0.6, 95% CI 2-sided [-0.77 to 1.95], Standard Error of Mean 0.69
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.712, MMRM; LS mean = 0.3, 95% CI 2-sided [-1.11 to 1.63], Standard Error of Mean 0.70
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.167, MMRM; LS mean = 1.0, 95% CI 2-sided [-0.41 to 2.38], Standard Error of Mean 0.71

14. Secondary Outcome: Change in MADRS Total Score From Randomization (Week 8) to Week 14
Description: as for outcome 1
Time Frame: Randomization (Week 8) to Week 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 159 | 149 | 131 | 164
units on a scale | -9.5 (0.59) | -10.6 (0.60) | -9.6 (0.62) | -11.0 (0.59)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization MADRS total score as a covariate. Treatment, visit and treatment by visit interaction are fixed effects the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.046, MMRM; LS mean = 1.5, 95% CI 2-sided [0.02 to 2.95], Standard Error of Mean 0.75
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.681, MMRM; LS mean = 0.3, 95% CI 2-sided [-1.17 to 1.79], Standard Error of Mean 0.75
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.087, MMRM; LS mean = 1.3, 95% CI 2-sided [-0.19 to 2.84], Standard Error of Mean 0.77

15. Secondary Outcome: Change in Functional Impairment From Randomization (Week 8) to End of Treatment (Week 16) as Measured by the Sheehan Disability Scale (SDS) Total Score
Description: Sheehan Disability Scale (SDS) is 5-item, self-administered scale that measures the extent a patient is impaired by their disease. Higher scores indicate more severe impairment. The SDS total score is calculated as the sum of the score for the 3 inter-correlated domains (school/work, social life, and family life/home responsibilities) and ranges from 0 (unimpaired) to 30 (highly impaired).
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 171 | 168 | 163 | 172
units on a scale | -6.08 (0.561) | -6.34 (0.569) | -6.21 (0.592) | -7.06 (0.556)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit, and treatment by visit interaction as explanatory variables and the randomization SDS total score as a covariate. Treatment, visit and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 1.000, MMRM — [p-value comment as in outcome 1, analysis 1]; LS mean = 0.98, 95% CI 2-sided [-0.464 to 2.427], Standard Error of Mean 0.736
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 1.000, MMRM — [p-value comment as in outcome 1, analysis 1]; LS mean = 0.72, 95% CI 2-sided [-0.740 to 2.188], Standard Error of Mean 0.746
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 1.000, MMRM — [p-value comment as in outcome 1, analysis 1]; LS mean = 0.85, 95% CI 2-sided [-0.649 to 2.346], Standard Error of Mean 0.762

16. Secondary Outcome: Change in Functional Impairment From Randomization (Week 8) to End of Treatment (Week 16) as Measured by SDS Work/School Domain Score
Description: A 5-item, self-administered scale that measures the extent a patient is impaired by their disease. Higher scores indicate more severe impairment. The 3 inter-correlated domains are school/work, social life, and family life/home responsibilities. The numerical rating for the work/school domain score is 0- 10, where 10 is considered to be 'highly impaired'.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 141 | 140 | 126 | 137
units on a scale | -2.0 (0.21) | -1.8 (0.22) | -1.9 (0.24) | -2.1 (0.22)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization SDS work/school domain score as a covariate. Treatment, visit and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.914, MMRM; LS mean = 0.0, 95% CI 2-sided [-0.54 to 0.61], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.446, MMRM; LS mean = 0.2, 95% CI 2-sided [-0.36 to 0.81], Standard Error of Mean 0.30
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.656, MMRM; LS mean = 0.1, 95% CI 2-sided [-0.47 to 0.75], Standard Error of Mean 0.31

17. Secondary Outcome: Change in Functional Impairment From Randomization (Week 8) to End of Treatment (Week 16) as Measured by SDS Social Life Domain Score
Description: A 5-item, self-administered scale that measures the extent a patient is impaired by their disease. Higher scores indicate more severe impairment. The 3 inter-correlated domains are school/work, social life, and family life/home responsibilities. The numerical rating for the SDS social life domain score is 0- 10, where 10 is considered to be 'highly impaired'.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 171 | 168 | 163 | 172
units on a scale | -2.1 (0.20) | -2.2 (0.20) | -2.2 (0.21) | -2.4 (0.20)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization SDS social life domain score. Treatment, visit and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.248, MMRM; LS mean = 0.3, 95% CI 2-sided [-0.21 to 0.82], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.498, MMRM; LS mean = 0.2, 95% CI 2-sided [-0.34 to 0.70], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.441, MMRM; LS mean = 0.2, 95% CI 2-sided [-0.32 to 0.74], Standard Error of Mean 0.27

18. Secondary Outcome: Change in Functional Impairment From Randomization (Week 8) to End of Treatment (Week 16) as Measured by SDS Family Life/Home Responsibilities Domain Score
Description: A 5-item, self-administered scale that measures the extent a patient is impaired by their disease. Higher scores indicate more severe impairment. The 3 inter-correlated domains are school/work, social life, and family life/home responsibilities. The numerical rating for the SDS family life/home responsibilities domain score is 0- 10, where 10 is considered to be 'highly impaired'.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 171 | 168 | 163 | 172
units on a scale | -2.0 (0.20) | -2.1 (0.20) | -2.0 (0.21) | -2.3 (0.20)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization SDS family life/home responsibilities domain score. Treatment, visit and treatment by visit interaction are effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.174, MMRM; LS mean = 0.4, 95% CI 2-sided [-0.16 to 0.87], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.402, MMRM; LS mean = 0.2, 95% CI 2-sided [-0.30 to 0.74], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.197, MMRM; LS mean = 0.3, 95% CI 2-sided [-0.18 to 0.88], Standard Error of Mean 0.27

19. Secondary Outcome: Change in Overall Quality of Life and Satisfaction From Randomization (Week 8) to End of Treatment (Week 16) by Assessing the Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) % Maximum Total Score
Description: The Q-LES-Q-SF (Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form) total score is derived by summing item scores 1 to 14. Higher scores are indicative of greater enjoyment or satisfaction in each domain. The Q-LES-Q-SF % maximum total score is calculated as 100% × (Q-LES-Q-SF total score - 14) / 56, and can range from 0% to 100%.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 171 | 166 | 162 | 172
units on a scale | 13.08 (1.388) | 13.24 (1.402) | 11.84 (1.409) | 14.55 (1.391)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; ANCOVA with randomization Q-LES-Q-SF % maximum total score as covariate, treatment as a fixed effect and pooled center as a random effect; Test type: Superiority or Other; p = 0.371, ANCOVA; LS mean = -1.47, 95% CI 2-sided [-4.697 to 1.756], Standard Error of Mean 1.643
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.432, ANCOVA; LS mean = -1.32, 95% CI 2-sided [-4.597 to 1.967], Standard Error of Mean 1.672
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.105, ANCOVA; LS mean = -2.71, 95% CI 2-sided [-5.992 to 0.573], Standard Error of Mean 1.672

20. Secondary Outcome: Change From Randomization (Week 8) to End of Treatment (Week 16) in Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q LES-Q-SF) Item 15
Description: The Q-LES-Q-SF (Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form) measures the patient's satisfaction with medication and overall quality of life. The 15th item queries respondents' satisfaction with the medication they are taking. Higher scores are indicative of greater enjoyment or satisfaction in each domain.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 153 | 154 | 151 | 157
units on a scale | 0.6 (0.08) | 0.7 (0.08) | 0.5 (0.08) | 0.7 (0.08)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; An analysis of covariance (ANCOVA) with randomization Q-LES-Q-SF item 15 score as covariate, treatment as a fixed effect and pooled center as a random effect; Test type: Superiority or Other; p = 0.312, ANCOVA; LS mean = -0.1, 95% CI 2-sided [-0.29 to 0.09], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.885, ANCOVA; LS mean = 0.0, 95% CI 2-sided [-0.18 to 0.21], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.067, ANCOVA; LS mean = -0.2, 95% CI 2-sided [-0.37 to 0.01], Standard Error of Mean 0.10

21. Secondary Outcome: Change From Randomization (Week 8) to End of Treatment (Week 16) in Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q LES-Q-SF) Item 16
Description: The Q-LES-Q-SF (Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form) measures the patient's satisfaction with medication and overall quality of life. The 16th item is a global rating of overall life satisfaction and contentment. Higher scores are indicative of greater enjoyment or satisfaction in each domain.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 170 | 166 | 162 | 172
units on a scale | 0.7 (0.08) | 0.7 (0.08) | 0.6 (0.08) | 0.8 (0.08)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; An analysis of covariance (ANCOVA) with randomization Q-LES-Q-SF item 16 as a fixed effect and pooled center as a random effect; Test type: Superiority or Other; p = 0.152, ANCOVA; LS mean = -0.1, 95% CI 2-sided [-0.33 to 0.05], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.078, ANCOVA; LS mean = -0.2, 95% CI 2-sided [-0.37 to 0.02], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.033, ANCOVA; LS mean = -0.2, 95% CI 2-sided [-0.41 to -0.02], Standard Error of Mean 0.10

22. Secondary Outcome: Change in EuroQol - 5 Dimensions (EQ-5D) From Randomization (Week 8) to End of Treatment (Week 16)
Description: A self-assessment questionnaire that provides 2 measures of health status. The EQ-5D index score is a weighted linear combination over 5 dimensions of health status. The score for each of the 5 dimensions can range from 1 to 3, and an equation is used to calculate the EQ-5D index score. The EQ-5D index score can range from possible negative values to a maximum of 1.0. The EQ-VAS is a visual analog scale with a range of 0 to 100. For both variables, a higher score indicates a better health state.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 171 | 168 | 163 | 172
units on a scale
  EQ-5D index score | 0.128 (0.0147) | 0.139 (0.0149) | 0.133 (0.0155) | 0.139 (0.0146)
  EQ-5D VAS score | 16.4 (1.52) | 17.0 (1.54) | 15.9 (1.61) | 18.7 (1.51)
Statistical Analysis 1: Comparison: 0.1 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization EQ-5D total score as a covariate. Treatment, visit and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.543, MMRM — Analysis for change in EQ-5D index score from randomization (Week 8) to end of treatment (Week 16); LS mean = -0.011, 95% CI 2-sided [-0.0465 to 0.0245], Standard Error of Mean 0.0181
Statistical Analysis 2: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Superiority or Other; p = 0.998, MMRM — Analysis for change in EQ-5D index score from randomization (Week 8) to end of treatment (Week 16); LS mean = 0.000, 95% CI 2-sided [-0.0360 to 0.0361], Standard Error of Mean 0.0183
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Superiority or Other; p = 0.743, MMRM — Analysis for change in EQ-5D index score from randomization (Week 8) to end of treatment (Week 16); LS mean = -0.006, 95% CI 2-sided [-0.0432 to 0.0308], Standard Error of Mean 0.0188
Statistical Analysis 4: Comparison: 0.1 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization EQ-5D VAS total score as a covariate. Treatment, visit and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.244, MMRM — Analysis of change in EQ-5D VAS score from randomization (Week 8) to end of treatment (Week 16); LS mean = -2.3, 95% CI 2-sided [-6.10 to 1.56], Standard Error of Mean 1.95
Statistical Analysis 5: Comparison: 1 mg BID TC-5214 vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Superiority or Other; p = 0.389, MMRM — Analysis of change in EQ-5D VAS score from randomization (Week 8) to end of treatment (Week 16); LS mean = -1.7, 95% CI 2-sided [-5.59 to 2.18], Standard Error of Mean 1.98
Statistical Analysis 6: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Superiority or Other; p = 0.165, MMRM — Analysis of change in EQ-5D VAS score from randomization (Week 8) to end of treatment (Week 16); LS mean = -2.8, 95% CI 2-sided [-6.79 to 1.16], Standard Error of Mean 2.02

ADVERSE EVENTS:
Groups:
- Placebo: Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + Placebo
Arm/Group | Placebo | 0.1 mg BID TC-5214 | 1 mg BID TC-5214 | 4 mg BID TC-5214
Serious Adverse Events (participants affected / at risk) | 2/174 | 2/174 | 4/174 | 2/171
Other Adverse Events (participants affected / at risk) | 64/174 | 68/174 | 72/174 | 94/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=174) | 0.1 mg BID TC-5214 (N=174) | 1 mg BID TC-5214 (N=174) | 4 mg BID TC-5214 (N=171)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=174) | 0.1 mg BID TC-5214 (N=174) | 1 mg BID TC-5214 (N=174) | 4 mg BID TC-5214 (N=171)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2) | 6 (6)
Constipation (Gastrointestinal disorders) | 11 (11) | 13 (13) | 13 (14) | 34 (35)
Dry Mouth (Gastrointestinal disorders) | 3 (4) | 5 (5) | 5 (5) | 18 (18)
Diarrhoea (Gastrointestinal disorders) | 12 (13) | 1 (1) | 3 (4) | 3 (4)
Nausea (Gastrointestinal disorders) | 9 (10) | 7 (8) | 6 (7) | 11 (11)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 5 (5)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (4) | 1 (1) | 4 (5) | 4 (4)
Fatigue (General disorders) | 4 (4) | 6 (6) | 10 (10) | 9 (9)
Influenza (Infections and infestations) | 8 (8) | 2 (2) | 6 (6) | 5 (5)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (4) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (2) | 5 (6)
Alanine Aminotransferase Increased (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 2 (3)
Increased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 23 (27) | 22 (27) | 24 (41) | 17 (17)
Dizziness (Nervous system disorders) | 7 (9) | 9 (9) | 13 (13) | 13 (14)
Somnolence (Nervous system disorders) | 5 (5) | 5 (5) | 7 (7) | 9 (10)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Insomnia (Psychiatric disorders) | 1 (1) | 6 (6) | 9 (11) | 7 (8)
Agitation (Psychiatric disorders) | 4 (4) | 3 (3) | 3 (3) | 5 (5)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Nightmare (Psychiatric disorders) | 2 (2) | 4 (4) | 1 (1) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 4 (4) | 7 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 8 (11)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
Hypertension (Vascular disorders) | 2 (2) | 2 (3) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days